CLINICAL TRIAL: NCT03583359
Title: Evaluation of Effectiveness and Safety of Radiesse (+) to Improve the Contour of Jawline by Adding Volume to the Jawline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M900391004
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Results first posted 2022-06-28 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Improvement of Jawline Contour

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment with Radiesse (+) (Experimental)
  Interventions: Device: Radiesse (+)
- Control/Delayed Treatment with Radiesse (+) (Other)
  Interventions: Device: Radiesse (+)

INTERVENTIONS:
Device: Radiesse (+) — Radiesse (+) for jawlines.
  Other Names: Radiesse (+) Injectable Dermal Filler with Lidocaine

SUMMARY:
To demonstrate the effectiveness and safety of Radiesse (+) following deep (subdermal and/or supraperiosteal) injection to improve the contour of jawline by adding volume to the jawline.

ELIGIBILITY:
Inclusion Criteria:

1. Has right and left jawline ratings of 2 or 3 (moderate or severe) on the Merz Jawline Assessment Scale (MJAS).
2. Has the same MJAS score on both jawlines (that is, jawlines are symmetrical).
3. Is greater than or equal to (>=) 22 and less than or equal to (<=) 65 years of age.

Exclusion Criteria:

1. Ever been treated with fat injections or permanent fillers (example, silicone, polymethylmethacrylate (PMMA)) in the lower face and/or jawline area or plans to receive such treatments during participation in the study.
2. Been treated with semi-permanent dermal fillers (example, poly L-lactic acid) in the lower face and/or jawline area in the past 5 years or plans to receive such treatments during participation in the study.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz North America, Inc.
Locations (15):
- United States (15):
  - Clinical Testing of Beverly Hills, Merz Investigational Site #0010395, Beverly Hills, California
  - Skin Care Center, Merz Investigational Site #0010099, Los Angeles, California
  - Ava MD, Merz Investigational Site #0010299, Santa Monica, California
  - Moradi MD Face Beautiful Inc, Merz Investigational Site #0010358, Vista, California
  - AboutSkin Research LLC, Merz Investigational Site #0010103, Greenwood Village, Colorado
  - Skin Research Institute, Merz Investigational Site #0010101, Coral Gables, Florida
  - Research Institute of the Southeast, LLC, Merz Investigational Site #0010420, West Palm Beach, Florida
  - Lupo Center for Aesthetic and General Dermatology, Merz Investigational Site #0010418, New Orleans, Louisiana
  - MD Laser Skin & Vein Institute, Merz Investigational Site #0010323, Hunt Valley, Maryland
  - SkinCare Physicians of Chestnut Hill. Merz Investigational #0010098, Chestnut Hill, Massachusetts
  - Skinfluence Medical PC, Merz Investigational #0010421, New York, New York
  - Bass Plastic Surgery PLLC, Merz Investigational Site #0010419, New York, New York
  - Dermatology, Laser & Vein Specialists of the Carolinas, Merz Investigational Site #0010194, Charlotte, North Carolina
  - Clinical Research Center of the Carolinas, Merz Investigational Site #0010417, Charleston, South Carolina
  - Westlake Dermatology, Merz Investigational Site #0010322, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moradi A, Green J, Cohen J, Joseph J, Dakovic R, Odena G, Verma A, Scher R. Effectiveness and Safety of Calcium Hydroxylapatite With Lidocaine for Improving Jawline Contour. J Drugs Dermatol. 2021 Nov 1;20(11):1231-1238. doi: 10.36849/jdd.6442. PMID 34784131
- [Derived] Moradi A, Dakovic R. Plain language summary of the pivotal study of calcium hydroxylapatite with lidocaine for improvement of jawline contour. J Dermatolog Treat. 2024 Dec;35(1):2421435. doi: 10.1080/09546634.2024.2421435. Epub 2024 Nov 6. PMID 39505354
- [Derived] Green JB, Del Campo R, Durkin AJ, Funt DK, Nasrallah N, Martinez K, Moradi A. Long-term duration and safety of Radiesse (+) for the treatment of jawline. J Cosmet Dermatol. 2024 Oct;23(10):3202-3209. doi: 10.1111/jocd.16436. Epub 2024 Jun 27. PMID 38934231

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15 investigational sites in the United States.
Pre-assignment Details: A total of 180 participants were enrolled and randomized in the study.
Groups:
- Treatment With Radiesse (+): Right and left jawline injected with Radiesse (+).
- Control/Delayed Treatment With Radiesse (+): Participants did not receive treatment for the first 12 weeks.
Period: Overall Study
Arm/Group | Treatment With Radiesse (+) | Control/Delayed Treatment With Radiesse (+)
Started | 123 | 57
Treated Participants | 122 | 53
Completed | 94 | 45
Not Completed | 29 | 12
Not completed — Withdrawal by Subject | 15 | 6
Not completed — Lost to Follow-up | 12 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population consisted of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment With Radiesse (+) | Control/Delayed Treatment With Radiesse (+) | Total
Number analyzed (Participants) | 123 | 57 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (7.3) | 55.0 (6.6) | 55.3 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 44 | 146
  Male | 21 | 13 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 9 | 31
  Not Hispanic or Latino | 101 | 48 | 149
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 10 | 24
  White | 103 | 42 | 145
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate According to the Merz Jawline Assessment Scale (MJAS)
Description: MJAS was a 5-point scale (0-4 scores; higher scores mean worse outcome). Responder rate was defined as percentage of participants with a greater than or equal to (>=) 1-point improvement.
Time Frame: At Week 12
Population: ITT population consisted of all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment With Radiesse (+) | Control/Delayed Treatment With Radiesse (+)
Number analyzed (Participants) | 123 | 57
percentage of participants | 75.6 [67.3 to 82.3] | 8.8 [3.8 to 18.9]
Statistical Analysis 1: Comparison: Treatment With Radiesse (+) vs Control/Delayed Treatment With Radiesse (+); Test type: Superiority; p < 0.0001, Fisher's exact test; The Fisher's exact test was utilized to test the superiority of treatment (Radiesse [+]) over control group; Difference in Responder Rate = 66.8, 95% CI 2-sided [53.7 to 75.2] — Two-sided Newcombe confidence intervals (CIs) were calculated for difference in responder rate

2. Primary Outcome: Number of Participants Reporting One or More Device and/or Injection Related Treatment-emergent Adverse Events (TEAEs) and Device and/or Injection Related Serious TEAEs
Time Frame: Baseline up to end of study (Week 60)
Population: The safety evaluation set (SES) was the subset of all participants who were exposed to study medication at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Radiesse (+) | Control/Delayed Treatment With Radiesse (+)
Number analyzed (Participants) | 122 | 53
Participants
  Participants with Device and/or Injection Related TEAEs | 36 | 10
  Participants with Device and/or Injection Related Serious TEAEs | 0 | 0

3. Secondary Outcome: Percent Change From Baseline in Face-Q Satisfaction
Description: The participant assessed satisfaction using the Face-Q Satisfaction with Lower Face and Jawline module (Rasch transformed score 0-100; higher scores mean better outcome).
Time Frame: Baseline up to Week 12
Population: ITT population consisted of all randomized participants. Here "overall number of participants analyzed" were participants who were evaluable for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Treatment With Radiesse (+) | Control/Delayed Treatment With Radiesse (+)
Number analyzed (Participants) | 115 | 53
percent change | 269.8 [215.1 to 324.6] | -9.4 [-28.2 to 9.5]

4. Secondary Outcome: Global Aesthetic Improvement Scale (GAIS) Scores as Assessed by the Treating Investigator
Description: GAIS ratings (-3 to +3 scores; lower scores mean worse outcome).
Time Frame: At Week 12
Population: ITT population consisted of all randomized participants. Here "overall number of participants analyzed" were participants who were evaluable for this outcome measure. As planned, this OM was evaluated only for participants in treatment with Radiesse (+) group.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Radiesse (+)
Number analyzed (Participants) | 116
Participants
  Very Much Improved | 37
  Much Improved | 51
  Improved | 27
  No Change | 1
  Worse | 0
  Much Worse | 0
  Very Much Worse | 0

5. Secondary Outcome: GAIS Scores as Assessed by Participants
Description: GAIS ratings (-3 to +3 scores; lower scores mean worse outcome).
Time Frame: At Week 12
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Radiesse (+)
Number analyzed (Participants) | 116
Participants
  Very Much Improved | 32
  Much Improved | 38
  Improved | 39
  No Change | 6
  Worse | 1
  Much Worse | 0
  Very Much Worse | 0

6. Secondary Outcome: Responder Rate According to the MJAS as Assessed by Independent Panel Reviewers (IPRs)
Description: MJAS was a 5-point scale (0-4 scores; higher scores mean worse outcome). Responder rate was defined as percentage of participants with a >=1-point improvement.
Time Frame: At Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment With Radiesse (+) | Control/Delayed Treatment With Radiesse (+)
Number analyzed (Participants) | 111 | 49
percentage of participants | 47.7 [38.7 to 57.0] | 8.2 [3.2 to 19.2]

ADVERSE EVENTS:
Time Frame: From first treatment up to the end of study (Week 60)
Description: The investigator reported AEs systematically at each visit.
Arm/Group | Treatment With Radiesse (+) | Control/Delayed Treatment With Radiesse (+)
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/53
Serious Adverse Events (participants affected / at risk) | 1/122 | 2/53
Other Adverse Events (participants affected / at risk) | 25/122 | 7/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With Radiesse (+) (N=122) | Control/Delayed Treatment With Radiesse (+) (N=53)
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With Radiesse (+) (N=122) | Control/Delayed Treatment With Radiesse (+) (N=53)
Injection site mass (General disorders) | 13 | 6
Injection site bruising (General disorders) | 11 | 1
Injection site pain (General disorders) | 8 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.

DOCUMENTS (2):
  • Study Protocol (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/59/NCT03583359/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/59/NCT03583359/SAP_001.pdf